CLINICAL TRIAL: NCT02093052
Title: Intervening Early With Neglected Children: Key Childhood Outcomes
Brief Title: Intervening Early With Neglected Children
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Mary Dozier, Principal Investigator, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIH R01 74374
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Conduct Disorder; ADHD; Depression
Keywords: Parenting; Parent child relations; Middle childhood outcomes
MeSH Terms: conditions — Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Attachment and Biobehavioral Catch-up (Experimental): Attachment and Biobehavioral Catch-up - 10 session intervention to enhance nurturance and following the lead
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up
- Developmental Education for Families (Active Comparator): Developmental Education for Families - 10 session intervention that targets cognitive development
  Interventions: Behavioral: Developmental Education for Families
- Low-risk (No Intervention): Low-risk comparison group

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up — Enhance nurturance and following the lead among parents. In-home intervention with parents and children present.
  Arms: Attachment and Biobehavioral Catch-up
Behavioral: Developmental Education for Families — Enhance children's cognitive development. In-home intervention with parents and children present.
  Arms: Developmental Education for Families

SUMMARY:
This study will assess early and middle childhood outcomes of an intervention for neglecting parents that was implemented in the children's infancy. We expect that parents who received the Attachment and Biobehavioral Catch-up Intervention in infancy will be more nurturing and will follow children's lead more than parents who received a control intervention, and that children will show better outcomes in attachment, inhibitory control, emotion regulation, and peer relations than children of parents who received the control intervention.

DETAILED DESCRIPTION:
Children were randomly assigned to receive the ABC intervention or a control intervention (DEF) in infancy. These two groups, plus a group of low-risk children, will be studied in early and middle childhood. Of interest will be differences in parent and child outcomes that result from the intervention.

Hypothesis 1: Neglected children whose parents received the ABC intervention and low-risk comparison children will show better inhibitory control than neglected children whose parents received the DEF intervention.

Hypothesis 2: Children in the ABC intervention condition and low-risk comparison children will show better emotion regulation than children in the DEF condition.

Hypothesis 3: Children in the ABC intervention condition and comparison children will show less reactive aggression and less hostile attributional bias than children in the DEF condition.

Hypothesis 4: Children in the ABC condition and comparison children will show more normative cortisol production than children in the DEF condition.

Although we expect that sustained changes in parenting are critical for sustained changes in child behaviors, several alternative models will be tested. First, it is possible that when parents change as a result of the intervention in a child's infancy, there are positive outcomes for children regardless of whether the changes in parenting are sustained. If this is the case, early parenting will mediate the effects of the intervention when controlling for later parenting. Second, if concurrent parenting is what is critical to child functioning, current parenting will mediate intervention effects on child outcomes when controlling for early parenting. Third, longitudinal modeling of both parent and child behaviors allows for analysis of cross-lagged associations using structural equation modeling. Such modeling can examine concurrent and transactional associations between parent and child. We can also examine associations between change at behavioral and biological levels.

Longitudinal modeling will be used to examine models of change in parenting behaviors and how those influence child outcomes.

ELIGIBILITY:
Inclusion Criteria:

* must have been in earlier randomized clinical trial

Exclusion Criteria:

-

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2005-03; Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Inhibitory control | Child age of 36 months
  DB-DOS- children who successfully do not touch forbidden toys
Emotion regulation | Child age of 36 months
  Children will complete emotion regulation tasks (Perfect Circle and Disappointing Gift)
Peer relations | Child age of 10 years
  Social information processing will be assessed through children's responses to videos of peer provocations.
Child diagnosis | Child age of 10
  Parents will complete diagnostic interview.
Child aggression | Child age of 10
  Children will complete video game that will allow assessment of reactive and proactive aggression.
Cortisol production | Child age of 24 months
  Salivary cortisol levels collected at wake-up and bedtime
Cortisol production | Child age of 8
  Salivary cortisol levels collected at wake-up and bedtime
Cortisol production | Child age of 10
  Salivary cortisol levels collected at wake-up and bedtime
Attachment | Age 18 months
  Attachment assessed through Strange Situation

SECONDARY OUTCOMES:
Parental sensitivity | Child age of infancy (12-24 months child age)
  Parental sensitivity will be assessed through parent-child interactions.
Child attachment security (narrative measure) | Child age 9
  Children's score on Attachment Script Assessment, a narrative technique
Child inhibitory control in middle childhood | Child age 8
  Delay task (Flanker). ERP data will be collected.
Autonomic nervous system activity | Child age 8
  Child heart rate and respiratory sinus arrhythmia
Child brain activity | Child age 9
  Child brain activation assessed in fMRI
Parent Attachment Script Knowledge | Child age of 9
  Parents' score on Attachment Script Assessment, a narrative technique
Parental sensitivity using Parent-Child Interaction Coding System | Child age 9
  Extent to which parent is responsive and attuned in support discussion (coded behaviorally)
Autonomic nervous system activity | Child age 10
  Child Respiratory Sinus Arrhythmia (RSA)
Alpha and theta wave | Child age 9
  Alpha and theta wave activity in resting state EEG
Round Robin Assessment of Peer Rejection | Child age 9
  Play groups of unknown peers constituted and video recorded; videos coded at microanalytic level for indices of peer rejection
Parent neural activity assessed through event related potentials | Child age 4
  Negative 170 ms. (N170: negative deflection 170 ms. after onset of stimulus) in task discriminating infant affect
Parent neural activity assessed through event related potentials | Child age 4
  Late positive potential - 350-600 ms after onset of stimulus (LPP) in task discriminating infant affect
Child attachment security (self-reported on Kerns' Attachment Inventory) | Child age 9
  Self-report from child of extent to which he or she can rely on parent
Child attachment security (self-reported on Kerns' Attachment Inventory) | Child age 10
  Self-report from child of extent to which he or she can rely on parent
Body mass index | Age 3
  Proportion of height to weight
Body mass index | Age 4
  Proportion of height to weight

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dozier, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Valadez EA, Tottenham N, Korom M, Tabachnick AR, Pine DS, Dozier M. A Randomized Controlled Trial of a Parenting Intervention During Infancy Alters Amygdala-Prefrontal Circuitry in Middle Childhood. J Am Acad Child Adolesc Psychiatry. 2024 Jan;63(1):29-38. doi: 10.1016/j.jaac.2023.06.015. Epub 2023 Jun 27. PMID 37385583
- [Derived] Hubbard JA, Bookhout MK, Zajac L, Moore CC, Dozier M. Children's social information processing predicts both their own and peers' conversational remarks. Dev Psychol. 2023 Jun;59(6):1153-1165. doi: 10.1037/dev0001510. Epub 2022 Dec 22. PMID 36548042
- [Derived] Garnett M, Bernard K, Hoye J, Zajac L, Dozier M. Parental sensitivity mediates the sustained effect of Attachment and Biobehavioral Catch-up on cortisol in middle childhood: A randomized clinical trial. Psychoneuroendocrinology. 2020 Nov;121:104809. doi: 10.1016/j.psyneuen.2020.104809. Epub 2020 Jul 24. PMID 32781397
- [Derived] Valadez EA, Tottenham N, Tabachnick AR, Dozier M. Early Parenting Intervention Effects on Brain Responses to Maternal Cues Among High-Risk Children. Am J Psychiatry. 2020 Sep 1;177(9):818-826. doi: 10.1176/appi.ajp.2020.20010011. Epub 2020 Jul 31. PMID 32731812
- [Derived] Zajac L, Raby KL, Dozier M. Sustained effects on attachment security in middle childhood: results from a randomized clinical trial of the Attachment and Biobehavioral Catch-up (ABC) intervention. J Child Psychol Psychiatry. 2020 Apr;61(4):417-424. doi: 10.1111/jcpp.13146. Epub 2019 Nov 1. PMID 31677152
- [Derived] Bernard K, Frost A, Jelinek C, Dozier M. Secure attachment predicts lower body mass index in young children with histories of child protective services involvement. Pediatr Obes. 2019 Jul;14(7):e12510. doi: 10.1111/ijpo.12510. Epub 2019 Jan 18. PMID 30659782
- [Derived] Bernard K, Hostinar CE, Dozier M. Intervention effects on diurnal cortisol rhythms of Child Protective Services-referred infants in early childhood: preschool follow-up results of a randomized clinical trial. JAMA Pediatr. 2015 Feb;169(2):112-9. doi: 10.1001/jamapediatrics.2014.2369. PMID 25436448

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02093052/Prot_SAP_000.pdf